CLINICAL TRIAL: NCT04189380
Title: Therapeutic Literacy Evaluation in Liver Transplanted Patients
Acronym: THELEHEPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RBHP 2018 TALAVERA; 2018-A01031-54 (Other: 2018-A01031-54)
Record Dates: First submitted 2019-11-28; First posted 2019-12-06 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Health Literacy; Liver Transplantation
Keywords: Health literacy; liver transplanted patients; cognitive evaluation; social status
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): liver transplanted patient
  Interventions: Other: HLQ (Health literacy questionnaire); Other: MoCA (Montreal Cognitive Assessment)

INTERVENTIONS:
Other: HLQ (Health literacy questionnaire) — each patient complete survey and self-assessment questionnaire before or after his medical consultation
Other: MoCA (Montreal Cognitive Assessment) — each patient complete survey and self-assessment questionnaire before or after his medical consultation

SUMMARY:
Health literacy is a new concept in therapeutic patient education. Health Literacy has been defined as the cognitive and social skills which determine the motivation and ability of individuals to gain access to, understand and use information in ways which promote and maintain good health. Health literacy seems predictive of adherence 's patients to treatment or positive health behavior.

Liver transplanted patients need to modify their lifestyle and to perform new behaviors in order to improve their survival and their quality of life. Health literacy evaluation in these patients is necessary to know what they understand and to improve their intake.

The Aim of the study is to evaluate health literacy among liver transplanted patient and to perform liver transplanted patient profiles related to their own health literacy.

The second aim is to study the impact of health literacy on medication adherence and iatrogenic hospitalizations It is a monocentric non-randomized study. During the hepatologist consultation, the HLQ Health Literacy Questionnaire is performed to explore patient health understanding and perception. Then the pharmacist interviews the patient to explore motivations and brakes for their own healthcare; Furthermore, a cognitive and precarity evaluation is performed in order to analyze psychological or social factors which can influence health literacy.

DETAILED DESCRIPTION:
Tests performed:

* Health Literacy Questionnaire: HLQ
* Montreal Cognitive Evaluation Assessment: MoCA
* EPICES: precarity test validated in French
* A qualitative interview

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 18 years
* Liver transplanted patient > 1 year at the start of the study
* patient who are followed-up by an hepatologist in the center
* patient who understands and speaks French

Exclusion Criteria:

* patient not yet liver transplanted (on the waiting-list)
* patient who has not come back home yet
* patient who does not speak or understand French
* patient refusal to participate
* patient under supervision or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
health literacy questionnaire | day 1
  a survey in 2 parts. Each part contains about twenty questions with Likert scale

SECONDARY OUTCOMES:
MoCA questionnaire | day 1
  evaluation of cognitive assessment and detection mild cognitive dysfunction at the consultation
EPICES questionnaire | day 1
  auto-evaluation of social and economic status

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Talavera, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France